CLINICAL TRIAL: NCT01534026
Title: Polypharmacy in the Heart Failure Patient: Are All Prescribed Drug Classes Required? Aspirin Withdrawal in Non-ischaemic Cardiomyopathy Study
Brief Title: Aspirin Withdrawal in Non-ischaemic Cardiomyopathy Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Dr Ingrid Hopper, The Alfred
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CP-01/12
Record Dates: First submitted 2012-02-02; First posted 2012-02-16 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Active Comparator): Current dose of aspirin for 12 weeks
  Interventions: Drug: Aspirin
- Withdrawal arm (Experimental): Withdrawal of aspirin for 12 weeks
  Interventions: Other: withdrawal of aspirin

INTERVENTIONS:
Drug: Aspirin — Current dose
  Arms: Aspirin
Other: withdrawal of aspirin — Stopping current dose of aspirin
  Arms: Withdrawal arm

SUMMARY:
Heart failure (cardiomyopathy) is a chronic condition in which the heart fails to function as a pump to move blood around the body. Aspirin has been traditionally used in heart failure because a tendency towards blood clots (including stroke and heart attack, clots in the legs and in the lungs) has been observed in this group and aspirin's mechanism of action is to prevent blood clots. This is important because two-thirds of cases of heart failure are caused by a blood clot in the coronary artery resulting in a heart attack, and aspirin is given to reduce the chances of further heart attacks.

However aspirin was introduced before clinical trials as the investigators know them now were run. Systematic review of the trials of aspirin in heart failure has shown that its use does not increase survival, and there is no evidence to recommend its routine use. Another important finding was that use of aspirin may reduce the beneficial effects of ACE inhibitors which do have a mortality benefit, and that aspirin was associated with an increase in hospitalisation for heart failure compared to other drugs which prevent clots or placebo.

The investigators propose that the use of aspirin in heart failure that is not caused by heart attacks ("non-ischaemic cardiomyopathy") is unnecessary and could be stopped. The importance of finding evidence to cease unproven medications in heart failure cannot be understated. Patients with heart failure take an average of six prescription medications each day. Each medication has side effects and the interactions of all the drugs together are unknown. Aspirin itself is a drug which frequently has side effects of increased risk of bleeding, gastrointestinal ulceration, as well as kidney impairment.

In this study, the investigators plan to withdraw aspirin from patients with stable non-ischaemic heart failure in a closely monitored environment and watch for the effect of this on heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years
2. In sinus rhythm at the time of randomisation
3. Have a LVEF <0.40
4. Are receiving ACE inhibitor or ARB, β-blocker and diuretic therapy at the optimal doses.
5. Has been receiving aspirin therapy for at least 3 months
6. Documented non-ischaemic heart failure. Must have at least 1 of the following:
7. Willing and able to provide informed consent

Exclusion Criteria:

1. Ischaemic cardiomyopathy
2. High risk of thromboembolism, including

   * atrial fibrillation
   * previous thromboembolic event including left ventricular thrombus, stroke or transient ischaemic attack, myocardial infarction, deep venous thrombosis or pulmonary embolus
   * an underlying condition which predisposes to thromboembolism e.g. amyloidosis
   * idiopathic dilated cardiomyopathy and a history of venous thromboembolism in a first degree relative
3. Systolic BP >160mmHg
4. Uncorrected primary valvular disease
5. Active myocarditis
6. Obstructive or restrictive cardiomyopathy
7. Exercise capacity limited by factors other than cardiac dyspnoea
8. Hospitalisation within one month of randomisation
9. Severe primary pulmonary (VC <1.5L), renal or hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in NYHA class | Week 12 and week 24
Change in 6 minute walk test | 12 week and 24 weeks
Change in BNP | 12 weeks and 24 weeks
change in Quality of Life questionnaire | 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia